CLINICAL TRIAL: NCT02923674
Title: Empowered With Movement to Prevent Obesity and Weight Regain
Acronym: EMPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Wake Forest University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00035300; R01AG051624 (NIH); R01AG051624-02S1 (NIH); R01AG051624-02S2 (NIH)
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Weight Loss; Sedentary Lifestyle
MeSH Terms: conditions — Obesity; Weight Loss; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight loss + sitless (Other): All participants will undergo a dietary WL intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass.
  Participants will be encouraged and taught to reduce sedentary behavior (SB) during waking hours. The SitLess treatment targets increases in postural shifts and light, spontaneous physical activity (SPA) (MET level <3).
  Interventions: Behavioral: Weight loss; Behavioral: Sitless
- Weight loss + exercise (Other): All participants will undergo a dietary WL intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass.
  Participants will be asked to perform structured aerobic exercise (mostly treadmill walking) of moderate-intensity for 4-5 days/week, progressing to a duration of 200 min/week.
  Interventions: Behavioral: Weight loss; Behavioral: Exercise
- Weight loss + exercise + sitless (Other): All participants will undergo a dietary WL intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass.
  Participants will be encouraged and taught to reduce sedentary behavior (SB) during waking hours. The SitLess treatment targets increases in postural shifts and light, spontaneous physical activity (SPA) (MET level <3).
  Participants will be asked to perform structured aerobic exercise (mostly treadmill walking) of moderate-intensity for 4-5 days/week, progressing to a duration of 200 min/week.
  Interventions: Behavioral: Weight loss; Behavioral: Exercise; Behavioral: Sitless

INTERVENTIONS:
Behavioral: Weight loss — All participants will undergo a dietary WL intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. The WL intervention includes nutrition education, state-of-the-art behavioral methods for promoting WL, and strategies that optimize self-regulation.
  Other Names: WL
Behavioral: Exercise — Perform structured aerobic exercise (mostly treadmill walking) of moderate-intensity for 4-5 days/week, progressing to a duration of 200 min/week. Participants will attend center-based sessions for at least 3 days/week during the first intensive 6-month phase and at least one day/week during the second 3-month transition phase (months 7-9), with recording of home-based exercise for the other 2-4 days/week.
  Other Names: EX
  Arms: Weight loss + exercise; Weight loss + exercise + sitless
Behavioral: Sitless — Encouraged and taught to reduce sedentary behavior (SB) during waking hours. The SitLess treatment targets increases in postural shifts and light, spontaneous physical activity (SPA) (MET level <3).
  Other Names: SL
  Arms: Weight loss + exercise + sitless; Weight loss + sitless

SUMMARY:
This study will help determine the appropriate type, amount and intensity of physical activity most beneficial for preventing weight regain after weight loss in older adults.

DETAILED DESCRIPTION:
The investigators will use a 3-group design in 180 older (65-85 years), obese (BMI=30-45 kg/m2), sedentary men and women, all of whom will undergo a 9-month Weight Loss (WL) intervention (6-mo intensive phase and 3-mo reduced contact phase), followed by a 9-month self-managed follow-up phase with minimal contact, to test our overall hypothesis that intervening on Sedentary Behavior (SitLess) will enhance long-term Weight Loss in this age group. The diet element of the intervention is identical across groups, but groups differ by activity intervention: 1) structured, moderate-intensity, aerobic exercise (EX) (WL+EX); 2) intervening on SB throughout the day (WL+SitLess); or 3) (WL+EX+SitLess).

ELIGIBILITY:
Inclusion Criteria:

* 65-85 years
* BMI=30-45 kg/m2
* Weight stable-no loss or gain (±5%) in past 6 mo
* Sedentary
* No contraindication for safe and optimal participation in exercise training
* Approved for participation by Medical Director
* Willing to provide informed consent
* Agree to all study procedures and assessments
* Able to provide own transportation to study visits and intervention

Exclusion Criteria:

* Dependent on cane or walker
* Reported unintentional or intentional weight loss or gain of >5% in past 6 mo Participation in regular resistance training and/or > 20 mins/day of aerobic exercise in past 6 months
* Cognitive impairment (MoCA score <22)
* Low bone density (T-score < -2.3 on hip or spine scan)
* Severe arthritis, or other musculoskeletal disorder
* Joint replacement or other orthopedic surgery in past 6 mos
* Joint replacement or other orthopedic surgery planned in next 2 years

  * Uncontrolled resting hypertension (>160/90 mmHg);
  * Current or recent past (within 1 year) severe symptomatic heart disease, uncontrolled angina, stroke, chronic respiratory disease other than asthma or COPD, any disease requiring oxygen use, neurological or hematological disease; cancer requiring treatment in past year, except non-melanoma skin cancers
  * Serious conduction disorder, new Q waves or ST-segment depression (>3 mm), or uncontrolled arrhythmia
  * Room air SpO2 (oxygen saturation) at rest or with exercise qualifying for supplementary oxygen (SpO2≤88%)
  * Abnormal kidney or liver function (2x upper limit of normal);
  * eGFR <45 mL/min/1.73m2
  * Anemia (Hb<13 g/dL in men/ <12 g/dL in women);
  * Uncontrolled diabetes (fasting glucose >140 mg/dl);
  * Deficient levels of vitamin D (25 hydroxyvitamin D level < 20 ng/mL) in those not taking a vitamin D supplement;
  * Smoker (No nicotine in past yr)
  * No heavy alcohol use (>14 drinks/week)
  * Unstable severe depression
* Regular use of: growth hormones, oral steroids, weight loss medications or prescription osteoporosis meds
* Current participation in other research study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Nicklas, PhD, Principal Investigator — Wake Forest University Health Sciences; W. Jack Rejeski, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest Baptist Health Sticht Center on Aging, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burdette JH, Laurienti PJ, Miron LL, Bahrami M, Simpson SL, Nicklas BJ, Fanning J, Rejeski WJ. Functional Brain Networks: Unique Patterns with Hedonic Appetite and Confidence to Resist Eating in Older Adults with Obesity. Obesity (Silver Spring). 2020 Dec;28(12):2379-2388. doi: 10.1002/oby.23004. Epub 2020 Nov 1. PMID 33135364
- [Derived] Fanning J, Opina MT, Leng I, Lyles MF, Nicklas BJ, Rejeski WJ. Empowered with Movement to Prevent Obesity & Weight Regain (EMPOWER): Design and methods. Contemp Clin Trials. 2018 Sep;72:35-42. doi: 10.1016/j.cct.2018.07.010. Epub 2018 Jul 17. PMID 30026128

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Weight Loss + Exercise + Sitless | Weight Loss + Exercise | Weight Loss + Sitless
Started | 60 | 60 | 63
Completed | 32 | 32 | 38
Not Completed | 28 | 28 | 25
Not completed — Clinic Closed Due to COVID-19 | 14 | 11 | 14
Not completed — Lost to Follow-up | 7 | 12 | 7
Not completed — Problem with intervention | 2 | 2 | 1
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Loss + Exercise + Sitless | Weight Loss + Sitless | Weight Loss + Exercise | Total
Number analyzed (Participants) | 60 | 63 | 60 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (4.0) | 69.6 (4.6) | 70.7 (4.1) | 70.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 48 | 141
  Male | 14 | 16 | 12 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 49 | 45 | 136
  Black | 18 | 14 | 15 | 47
Region of Enrollment [Number; unit: participants]
  United States | 60 | 63 | 60 | 183
Education (>High School) [Count of Participants; unit: Participants] | 57 | 49 | 52 | 158
Cognitive Status (MoCA) Score [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment (MoCA) is to help determine if impaired cognition would preclude them from participating. The test is administered in approximately 10 minutes and it assesses several cognitive domains. Scores range from 0 to 30, with a lower score indicating cognitive impairment.
  units on a scale | 26.2 (2.3) | 26.1 (2.2) | 25.3 (2.2) | 25.86 (2.27)
Depression (CES-D) Score [Mean (Standard Deviation); unit: units on a scale] — Center for Epidemiological Studies-Depression (CES-D) is administered to help exclude potential participants with clinically significant depression. The CES-D is a 20-item tool that asks subjects to rate how often over the past week they experienced symptoms associated with depression. Scores range from 0 to 60, with high scores indicating greater depressive symptoms. A cutoff score of 16 or greater is indicative of clinical depression.
  units on a scale | 6.4 (5.1) | 6.0 (5.2) | 6.48 (6.4) | 6.31 (5.57)
Height [Mean (Standard Deviation); unit: cm] | 165.0 (7.5) | 165.4 (9.3) | 162.2 (8.9) | 164.3 (8.6)
Body Mass [Mean (Standard Deviation); unit: kg] | 96.8 (12.8) | 97.2 (14.3) | 94.3 (14.0) | 95.8 (13.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.4 (3.7) | 35.4 (3.8) | 35.5 (3.8) | 35.4 (3.8)
Waist to Hip Ratio [Mean (Standard Deviation); unit: ratio] — A score is calculated by dividing waist circumference by hip circumference. High risk for men is a score greater than or equal to 0.95 and greater than or equal to 0.86 for women.
  ratio | 0.88 (0.10) | 0.90 (0.09) | 0.88 (0.10) | 0.9 (0.3)
Gait Speed [Mean (Standard Deviation); unit: m/sec] | 1.00 (0.17) | 1.03 (0.19) | 1.00 (0.16) | 1.0 (0.2)
Short Physical Performance Battery (SPPB) Score [Mean (Standard Deviation); unit: units on a scale] — The SPPB consists of a test of balance, gait speed test, and chair stand, performed in this order to measure lower-extremity function. A score is totaled and can equal 0 to 12 with a lower score indicating poorer mobility and physical function.
  units on a scale | 10.8 (1.1) | 10.5 (1.4) | 10.7 (1.4) | 10.7 (1.3)
Expanded Short Physical Performance Battery (eSPPB) Score [Mean (Standard Deviation); unit: units on a scale] — Consists of a test of balance, gait speed test, and chair stand, performed in this order. The following equipment is required for the expanded SPPB: digital stopwatch, masking tape, measuring tape, script, and a straight-backed armless chair with a hard seat. To eliminate the effect of different footwear on test performance, tests are performed in tennis shoes or comfortable walking shoes with minimal or no heels. Tests are individually scored 0-4 and then totaled for a maximal score of 12. The higher a score, the better an individual's mobility and functional ability.
  units on a scale | 2.2 (0.3) | 2.2 (0.4) | 2.3 (0.3) | 2.2 (0.3)
Aerobic fitness [Mean (Standard Deviation); unit: VO2peak; ml/kg/min] — Measured during a maximal graded exercise test (GXT) to exhaustion on a treadmill using a RAMP protocol. The GXT is used to rule out any latent coronary artery disease and to measure cardiovascular functional capacity and peak oxygen uptake. The speed is set at the fastest speed that the participant can maintain for several minutes, and the grade steadily increases until the test is stopped. The respiratory rate, minute ventilation, breathing reserve, VO2, VCO2, respiratory exchange ratio, MET level, HR, VO2/HR, Kcal/min, RPE and BP at test conclusion are recorded.
  VO2peak; ml/kg/min | 22.2 (4.8) | 20.3 (5.0) | 21.2 (3.9) | 20.6 (4.1)
Resting Seated Blood Pressure--Systolic [Mean (Standard Deviation); unit: mmHg] | 132 (13) | 135 (12) | 135 (13) | 134.8 (14.2)
Resting Seated Blood Pressure Diastolic [Mean (Standard Deviation); unit: mmHg] | 82 (8) | 81 (8) | 82 (7) | 82 (8.9)
Self-reported comorbidity Hypertension [Count of Participants; unit: Participants] | 40 | 36 | 43 | 119
Self-reported comorbidity Diabetes [Count of Participants; unit: Participants] | 7 | 11 | 5 | 23
Self-reported comorbidity Sleep Apnea [Count of Participants; unit: Participants] | 24 | 19 | 19 | 62
Self-reported comorbidity Osteoarthritis [Count of Participants; unit: Participants] | 42 | 43 | 43 | 128
Self-reported comorbidity Osteopenia [Count of Participants; unit: Participants] | 14 | 9 | 15 | 38
Anti-hypertensive Medication use [Count of Participants; unit: Participants] | 42 | 41 | 44 | 127
Cholesterol-lowering Medication use [Count of Participants; unit: Participants] | 32 | 30 | 33 | 95
Glucose control Medication use [Count of Participants; unit: Participants] | 6 | 11 | 4 | 21
Anti-depressant/mood Medication use [Count of Participants; unit: Participants] | 16 | 16 | 20 | 52

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Measured in clinic on the same scale
Time Frame: Baseline
Population: The CONSORT represents all 6 waves while our results only include data for Waves 1-4 due to COVID restrictions impacting the 18mo visit data for Waves 5 and 6.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Weight Loss + Exercise + Sitless | Weight Loss + Exercise | Weight Loss + Sitless
Number analyzed (Participants) | 26 | 31 | 31
kg | 94.7 (10.2) | 91.6 (14.3) | 95.1 (14.3)

2. Primary Outcome: Body Weight
Description: Measured in clinic on the same scale
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Weight Loss + Exercise + Sitless | Weight Loss + Exercise | Weight Loss + Sitless
Number analyzed (Participants) | 26 | 31 | 33
kg | 86.9 (12.4) | 82.8 (11.4) | 87.0 (13.3)

3. Primary Outcome: Body Weight
Description: Measured in clinic on the same scale
Time Frame: 18 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Weight Loss + Exercise + Sitless | Weight Loss + Exercise | Weight Loss + Sitless
Number analyzed (Participants) | 26 | 31 | 33
kg | 89.8 (14.3) | 87.2 (13.1) | 88.7 (14.3)

4. Other Pre Specified Outcome: Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale
Description: 13 item scale used to measure fatigue over the past week with a 4-point Likert scale. The score range is 0-52 with a score of less than 30 indicating severe fatigue, and higher score denoting a better quality of life.
Time Frame: Baseline (0mo), 6mo, 18mo
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form 8a
Description: DAn 8 item questionnaire that assess fatigue over the past 7 days. All items are summed with the lowest possible score equaling 8 and the highest, a 40. A higher score indicates more fatigue.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Pittsburg Fatigability Questionnaire
Description: 10 item scale that assesses fatigability (fatigue in the context of a standardized task). A higher score indicates a higher performance fatigability, slower gait speed, worsening physical function.
  A 10 item scale that assesses fatigability (fatigue in the context of a standardized task). Score range is 0-50 with a higher score = a higher performance fatigability, slower gait speed, worsening physical function.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Short Form 36 Item (SF-36) Health Survey
Description: A 36 item survey of overall health broken into 8 scaled scores of vitality, physical function, pain, general health, mental health, social, physical, and emotional role functioning. Ranging from 0 to 100, the lower a person scores, the more disability.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Self-Efficacy for Walking Scale
Description: Self-reported measure used to determine a person's belief in their physical capability to successfully complete incremental walking distances (5-40 minutes) at a moderate pace. The total strength for each measure of self-efficacy is then calculated by summing the confidence ratings and dividing by the total number of items in the scale, resulting in a maximum possible efficacy score of 100.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Satisfaction With Physical Function Questionnaire
Description: A scale testing how satisfied an individual is with their physical fitness and abilities. Levels of satisfaction are rated on a 7 point scale from very dissatisfied to very satisfied. All items are then averaged to create a score ranging from -3 to 3.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Self-Efficacy for Managing Eating Questionnaire
Description: Used to measure self-efficacy for appropriate eating using 5 subscales (Negative Emotions, Availability, Social Pressure, Physical Discomfort, Positive Activities) of 4 items each (e.g., "I can resist eating even when high-calorie foods are available"). Item responses range from 0 (not confident) to 9 (very confident). An average score is created for each subscale and then a total score by averaging across all items. On a scale from 10 to 40, higher scores represent greater confidence in being able to restrain oneself from eating under difference contexts.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Experiences in Close Relationships Questionnaire
Description: Scale used to evaluate the construct of adult attachment by examining avoidance and anxiety. A person rates each statement about connection using a 7-point Likert scale which ranges from 1 (strongly disagree) to 7 (strongly agree). To obtain score, average responses from all 36 items. A score will range from 7 to 42 with a higher score representing insecure attachment.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Mindful Attention Awareness Scale (MAAS)
Description: 15-item questionnaire used to assess the core characteristic of mindfulness, or an awareness of and attention to what is taking place in the present. The 15 items are collected in a Likert scale, totaled, and averaged for a final score ranging from 1-7. A higher score reflects higher levels of mindfulness and a lower score is indicative of a negative emotional state.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Power of Food Questionnaire
Description: Scale assessing the psychological impact of living in food-abundant environments. It measures appetite for, rather than consumption of, palatable foods, at three levels of food proximity (food available, food present, and food tasted).
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Perceived Stress Scale
Description: A questionnaire used to measure the perception of stress and how often a person felt that way in the last month. Individual scores range from 0 to 40 with higher scores indicating a person perceives higher levels of stress which could lead to or correlate with negative behaviors such as stress eating or decreases in physical activity
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Food Cravings Questionnaire
Description: 15-item measure of short-term changes in food cravings. Responses are made on a five-point Likert scale with response categories ranging from 1 (strongly disagree) to 5 (strongly agree). The scale yields a sum total from the five subscale scores, including, 1) an intense desire to eat; 2) anticipation of positive reinforcement that may result from eating; 3) anticipation of relief from negative states and feelings as a result of eating; 4) obsessive preoccupation with food or lack of control over eating; and 5) craving as a physiological state. Sum scores range from 15 to 90 with higher scores representing more frequent and intense experiences of craving food.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Technology Survey
Description: Administered during assessment visits to gain insight on the participants' opinion of the technology (i.e., Empower application and web-based questionnaires, any tests/emails received from the Empower team) used in the study. Examples of these open-ended questions include: 1) How useful did you find the Empower smartphone app?; 2) To what extent was the Empower app a burden to use?; 3) How difficult or easy was the app to use?; 4) How important did you feel the app was to your experience in the Empower study?; 5) What were one or two of your favorite and least favorite features of the Empower app? Questions were not scored or used in data analysis, but provided staff with an overall user opinion as well as constructive criticism in order to improve similar technologies in future studies.
Time Frame: 6mo, 18mo
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Intervention Survey
Description: Administered at assessment visits to gain inside on the participants' opinion on the group dynamic used in the first 6 months of the study. Examples of the dichotomous questions include: 1) Did you enjoy working with the staff and participants?; 2) Did you feel pressured by staff and or participants to do well in the study?; 3) Did you get along with the staff and participants in Empower?; 4) Did you feel comfortable expressing your ideas and opinions to staff members and fellow participants?; 5) Do you feel people a part of the Empower study care about you? Questions were not scored or used in data analysis, but provided staff with an overall opinion of participant experience as well as constructive criticism in order to improve similar group settings in future studies.
Time Frame: 6 mo, 18 mo
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Anthropometric Measures
Description: Three anthropometric measures at three anatomical locations are taken using a handheld measuring table with tension and recorded in centimeters. The waist measurement is taken at the narrowest part of the torso below the ribcage and above the umbilicus. The hip measurement is measured at the maximal circumference of the buttocks. The mid-thigh is taken with the knee bent to 90°, midway between the inguinal crease and the proximal border of the patella. The measurements taken at each site are averaged. A waist/hip ratio is calculated.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Expanded Short Physical Performance Battery (eSPPB)
Description: Consists of a test of balance, gait speed test, and chair stand, performed in this order. The following equipment is required for the expanded SPPB: digital stopwatch, masking tape, measuring tape, script, and a straight-backed armless chair with a hard seat. To eliminate the effect of different footwear on test performance, tests are performed in tennis shoes or comfortable walking shoes with minimal or no heels. Tests are individually scored 0-4 and then totaled for a maximal score of 12. The higher a score, the better an individual's mobility and functional ability.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Treadmill Fatigability
Description: Test is done on a treadmill to assess perceived fatigability at a given workload. Participants are asked to rate their RPE (rating of perceived exertion) just as they start walking (0 min, 2.0 mph), half way through (2.5 min, 2.0 mph), and at the end of the test (5 min, 2.0 mph). Heart rate via a heart rate monitoring watch will be recorded at these same intervals.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Peak Aerobic Capacity (VO2) Peak
Description: Measured during a maximal graded exercise test (GXT) to exhaustion on a treadmill using a Raise, Activate, Mobilise, Potentiate (RAMP) protocol. The GXT is used to rule out any latent coronary artery disease and to measure cardiovascular functional capacity and peak oxygen uptake. The respiratory rate, minute ventilation, breathing reserve, VO2, Validation of Carbon Dioxide Production (VCO2), respiratory exchange ratio, one metabolic equivalent (MET) level, heart rate (HR), VO2/HR, kilocalorie/minutes (Kcal/min), Rating of Perceived Exertion (RPE) and Blood pressure (BP) at test conclusion are recorded.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Grip Strength
Description: The Jaymar Handheld Dynamometer is used to measure grip strength in both hands. To the nearest and highest kilogram achieved, hand grip strength is a commonly used measure of upper body skeletal muscle function and has been widely used as a general indicator of frailty with predictive validity for both mortality and functional limitation.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Resting Metabolic Rate (RMR)
Description: A facemask will be placed on the participant while he/she is lying on the exam table. Measures of oxygen consumption and carbon dioxide production will be collected continuously for 30 minutes and the RMR will be calculated using the Weir equation.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Activity Monitor
Description: Used to evaluate time spent in sedentary behavior, light, and moderate to vigorous physical activity (MVPA). An activPAL™ accelerometer (PAL Technologies, Glasgow, Scotland) is worn for 7-days at each of the three assessment visits: baseline, 6-months and 18-months. The monitor uses accelerometer-derived information about thigh position to estimate time spent in different body positions: lying or sitting = sedentary; standing still; and stepping = light and MVPA. Data is downloaded at the end of each 7-day period and cleaned and summarized for statistical analyses. The proprietary algorithm in the activPAL software is used to generate estimates of (a) Total Daily Energy Expenditure (TDEE); (b) sedentary time during the day, (c) number of breaks in sedentary time, (d) minutes spent in light activity, and (e) number of minutes spent in MVPA.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Ecological Momentary Assessment (EMA)
Description: Used to determine the relationship between dynamic food variables, physical activity variables, and long-term weight loss. Prior to the start of the intervention and following the initial intervention period, participants complete week-long daily assessments. The following are the different scales and questions asked of participants: 1) Affective Valence from the Feelings Scale (scored 0 - 10 where 0 = very bad and 10 = very good). 2) Six items from the exercise-induced feelings inventory, each on a 0 ="do not feel" to 10="feel very strongly" score. Calm, peaceful, and relaxed are then averaged for a "tranquility" subscale; "fatigued, "tired" and "worn-out" are averaged for a physical exhaustion subscale. 3) Hunger was queried by "How hungry are you right now?" where 0 = not at all hungry, and 10 = very hungry. 4) An individual's craving for food was queried by "How much do you crave eating your favorite food or snack right now?" where 0 = "do not feel" and 10 = "feel very strongly".
Time Frame: Baseline, 6mo
Reporting Status: Not Posted

26. Other Pre Specified Outcome: 400 Meter Walk Test
Description: Test is completed at a quick pace (without running) that the participant can maintain over the flat, 400 meter course. Timing begins when the participant takes his/her first step. Timing ends when the participant's whole foot crosses the line at the end of the 10th lap or the participant requests to stop. Recorded is the distance completed and time walked in minutes and seconds.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Walking Efficiency
Description: Used to determine the number of calories burned while walking at 2.0 mph on a treadmill with zero grade. Heart rate (HR) is measured continuously using a heart rate monitoring watch and will be recorded every minute. Blood pressure (BP) is monitored and recorded every minute. The test is terminated when the (HR) remains at a steady state (is within 5 beats per minute of the HR from the previous minute). The time to achieve steady state heart rate, the respiratory rate, minute ventilation, breathing reserve, VO2, VCO2, respiratory exchange ratio, MET level, HR, VO2/HR, Kcal/min, and the BP at steady state are recorded.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Visceral Fat
Description: A visceral fat measurement is obtained through a dual-energy X-ray absorptiometry (DEXA) whole body scan in a 5-cm wide region across the entire abdomen just above the iliac crest at a level approximate with the 4th lumbar vertebrae. Mass visceral fat is measured to the nearest gram and volume to the nearest centimeter.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Bone Mineral Density (BMD)
Description: Hip and spine BMD is measured using specific scans of the anterior-posterior spine Lumbar vertebrae 1-Lumbar vertebrae 4 (L1-L4) and proximal femur by dual-energy X-ray absorptiometry. BMD is recorded as a t-score with a lower score indicative of less bone density and increased risk for osteoporosis.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Cardiometabolic Risk Factors--Lab Work
Description: An 8-hour fasting venous blood sample is collected to measure cardiometabolic changes lipoprotein lipids, C-reactive protein, HbA1c, glucose and insulin.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Satisfaction With Physical Function
Description: Scale used to test how satisfied participants are with their physical fitness, functional ability, and physical appearance. Participants rate their level of satisfaction on a 7-point scale from very dissatisfied to very satisfied. Average all items to create a score ranging from -3 to 3. Higher values represent greater satisfaction with physical function and importance.
Time Frame: Baseline, 6mo, 18mo
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through month 18
Arm/Group | Weight Loss + Exercise + Sitless | Weight Loss + Sitless | Weight Loss + Exercise
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/63 | 0/60
Serious Adverse Events (participants affected / at risk) | 8/60 | 7/63 | 4/60
Other Adverse Events (participants affected / at risk) | 39/60 | 26/63 | 25/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss + Exercise + Sitless (N=60) | Weight Loss + Sitless (N=63) | Weight Loss + Exercise (N=60)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Takatsubu cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Complication of laparoscopic banding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Post Viral Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery bypass graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Gastric sleeve procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Knee replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Brain aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal benign mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss + Exercise + Sitless (N=60) | Weight Loss + Sitless (N=63) | Weight Loss + Exercise (N=60)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Takatsubu cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Capsulitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Achilles tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Knee sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
TMJ pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental Crown Replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcerative colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (3) | 2 (2) | 1 (1)
Bronchial infection (Infections and infestations) | 5 (6) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (3)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacterial gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (fungal) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (5) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (5) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Complication of laparoscopic banding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Car/Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Car/Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vaccine reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Medication Side Effect (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Retro-peritoneal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stenosis of branch of left middle cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Light headed (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Post viral neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 2 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eustachian tube infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
cataracts (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
retinal vascular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hip replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Bilateral blepharoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cataract surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cataract surgery (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
Coronary artery bypass graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Epidural injection (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Excision of skin cancers (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Gastric sleeve procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Joint injection (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Saphenous vein ablation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Phlebotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Knee replacement (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Achilles tendon repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Removal of ingrown toe nail (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Brain aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gallbladder pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal benign mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT02923674/Prot_SAP_002.pdf
  • Informed Consent Form (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT02923674/ICF_001.pdf